CLINICAL TRIAL: NCT01264159
Title: Preemptive Lung Impedance-guided Therapy of Evolving Acute Heart Failure in Acute Myocardial Infarction Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The principle investigator decided to change the protocol
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0090-10-HYMC
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Acute Heart Failure
Keywords: Developing acute heart failure

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Other: Usual treatment of patients with developing acute heart failure
- Lung impedence-guided treatment (Active Comparator)
  Interventions: Device: Lung impedence-guided therapy

INTERVENTIONS:
Device: Lung impedence-guided therapy
  Arms: Lung impedence-guided treatment
Other: Usual treatment of patients with developing acute heart failure
  Arms: Control

SUMMARY:
It is well known that 20-25% of patients hospitalized for acute myocardial infarction will develop acute heart failure during their hospitalization. Currently, the investigators have no reliable parameter for prediction of evolving acute heart failure in such a group of patients. As a result, the investigators have no way of preventing acute heart failure. Treatment of these patients only begins after appearance of clinical signs of acute heart failure. Lung impedance monitoring may be a good non-invasive parameter for prediction of evolving acute heart failure. This study will attempt to address whether preemptive lung impedence-guided therapy may prevent the development of overt acute heart failure and improve their clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the ICCU for acute myocardial infarction and developing acute heart failure during their hospitalization

Exclusion Criteria:

* Patients with acute myocardial infarction with clinical and radiological signs of acute heart failure at admission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Prevention of acute heart failure development in acute MI patients | Three years

SECONDARY OUTCOMES:
Improvement of clinical outcome in patients with lung impedence-guided treatments | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel